CLINICAL TRIAL: NCT07034274
Title: National Tunisian Clinical Registry on CardioVascular Secondary Prevention Clinical
Acronym: NATURE STOP-CH
Status: Recruiting | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Tunisian Society of Cardiology and Cardiovascular Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: DAC-017-NATURE STOP-CHD
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Secondary Prevention; CHD; CV Risk
Keywords: Secondary Prevention; STCCCV; CHD; CV Risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Event: Patient with any coronary event

SUMMARY:
A non-interventional, national longitudinal multicenter study of CV secondary prevention in Tunisia

DETAILED DESCRIPTION:
The NATURE-STOP-CHD study is carried out in Tunisia at cardiology consultations in hospitals and in the liberal sector. The study is a longitudinal non-interventional registry of patient undergoing secondary CV prevention. The data collected are managed by the DACIMA Clinical Suite® platform, which complies with international standards: FDA 21 CFR part 11 (Food and Drug Administration 21 Code of Federal Regulations part 11), HIPPA (Health Insurance Portability and Accountability Act), ICH (International Conference on Harmonisation), MedDRA (Medical Dictionary for Regulatory Activities). The DACIMA Clinical Suite® platform allows to track the data entered, check for inconsistencies and missing data, and schedule monitoring visits. A Steering Committee is set up to monitor patient inclusions, verify data sources, perform audit trails and prepare the statistical analysis plan for the study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 80 years
* Patients who have been hospitalized for at least one acute coronary event with coronary revascularization, either percutaneous or surgical by coronary artery bypass grafting, or who have confirmed coronary artery disease requiring optimal medical treatment for more than 6 months
* Coronary event happening in 2024
* Informed, read and signed consent

Exclusion Criteria:

* Familial hypercholesterolemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had a coronary event in 2024
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Compliance | From enrollment to the end of the follow-up (12 months)
  Number of subjects with sufficient adherence to their cardiovascular medication

CONTACTS AND LOCATIONS:
Overall Officials: Youssef Ben Ameur, MD, Study Chair — Tunisian Society of Cardiology and Cardiovascular Surgery; Salma Charfeddine, MD, Study Chair — Tunisian Society of Cardiology and Cardiovascular Surgery; Ihsen Zairi, MD, Study Chair — Tunisian Society of Cardiology and Cardiovascular Surgery
Locations (1):
- Tunisian Society of Cardiology and Cardiovascular Surgery, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
Needs prior authorization from the National Authority for the Protection of Personal Data, for any health data transfer outside the Tunisian territory

REFERENCES:
- See also: Website of the Tunisian Society of Cardiology and Cardiovascular Syrgery — https://stcccv.org.tn/